CLINICAL TRIAL: NCT03416400
Title: Characterization of a Method of Fertility Preservation for Patients Diagnosed for a Cancer
Brief Title: Comparison of Vitrification Effect Before or After In Vitro Maturation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Origio A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: CHU-372
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Oocytes Vitrified at Prophase-I Stage; Oocytes Matured in Vitro
Keywords: Vitrification; In vitro maturation; Cytoskeleton; chromosomes; High resolution imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Immature oocytes vitrified before In Vitro Maturation: Immature oocytes were vitrified using closed system vitrification. After warming, they were cultured during 36 hours in IVM medium and fixed for cellular analysis
  Interventions: Other: Oocyte vitrification
- Immature oocytes cultured in vitro before vitrification: Immature oocytes were cultured in vitro in IVM medium during 36 hours. After IVM, they were vitrified. After warming, they were fixed for cellular analysis.
  Interventions: Other: Oocyte vitrification
- Fresh oocytes: Immature oocytes were cultured in vitro in IVM medium during 36 hours and subsequently, fixed for cellular analysis.
  Interventions: Other: Oocyte vitrification

INTERVENTIONS:
Other: Oocyte vitrification — Immature oocytes were collected from patients (≤37 years old, without endometriosis, Polycystic syndrome or other ovulatory desease) who underwent to ICSI. In addition, immature oocytes collected from patient diagnosed with cancer will be included in this study. Oocytes were matured in vitro with IVM medium and vitrified in closed system (Vitrolife). Kinetic of maturation were analyzed by Primovision (Vitrolife) and actin, and spindle organization were studied by microscopy, immunostaining techniques and quantitive analysis.

SUMMARY:
Human oocyte cryopreservation is routinely used for fertility preservation of women who will be exposed to gonadotoxic effect of cancer treatment. After ovarian stimulation, matured oocytes are vitrified. However, this strategy cannot always be used, particularly for hormone-sensitive cancer or when ovarian stimulation is not possible. An approach including immature oocytes and in vitro maturation (IVM) could be considered in these cases. While some qualitative analysis of oocytes vitrified before or after IVM suggest that vitrification should be performed after IVM, little is known about vitrification effects on actin and tubulin cytoskeleton and kinetic of maturation of human ovocytes.

To answer to this question, Investigator performed quantitive analyses comparing matured oocytes from three different groups: vitrified before IVM or after IVM and non-vitrified oocytes. Non-vitrified matured oocytes were used as a control. Different parameters have been analysed during maturation and in matured oocytes.

DETAILED DESCRIPTION:
Immature oocytes were collected from patients (≤37 years old, without endometriosis, Polycystic syndrome or other ovulatory desease) who underwent to ICSI. In addition, immature oocytes collected from patient diagnosed with cancer will be included in this study. Oocytes were matured in vitro with IVM medium and vitrified in closed system ("Vitrolife"). Kinetic of maturation were analyzed by Primovision ("Vitrolife") and actin, and spindle organization were studied by microscopy, immunostaining techniques and quantitive analysis.

ELIGIBILITY:
Inclusion Criteria:

* - ICSI treatment
* Immature oocytes
* < 37 years old

Exclusion Criteria:

* - Polyckistic Ovarian Syndrome
* Endometriosis
* Ovulatory disease

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: female
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Analysis of maturation kinetic of oocytes vitrified at Prophase-I stage compared to fresh oocytes | at day 1
  After oocytes retrieval, immature oocytes will be vitrified (Rapid Vit Ovocyte®, Vitrolife) in a closed system (Rapid-I®, Vitrolife) and thawed for in vitro maturation few days after. The meiotic process will be analyzed by time lapse technology (Primovision®, Vitrolife). This will permit to score the time of maturation from resumption to polar body extrusion of ovocytes.

SECONDARY OUTCOMES:
Analysis of actin and tubulin cytoskeleton at Metaphase-II stage | at day 1
  Metaphase-II stage oocytes from both protocols will be used for Immuno-Fluorescence experiments to stain actin, tubulin and chromosomes. Oocytes will be imaged using confocal microscope to perform high resolution imaging and quantitative image analysis. The length, position and orientation of the second meiotic spindle will be quantifying. The actin network and chromosomes will be analyzed quantitatively. All measurements will be compared with fresh Metaphase-II oocytes used as a control group.
Analysis of chromosome segregation during the first meiotic division. | at day 1
  The first asymmetric division is highly error prone. To investigate whether chromosomes are segregated accurately after vitrification, we will perform Fluorescence In Situ Hybridization to paint each chromosome after chromosome spread from Metaphase-II stage oocytes from both conditions
Analysis of cortical granules distribution in Metaphase-II stage oocytes. | at day 1
  A staining with Lectin will be used to mark cortical granules of matured oocytes from both protocols to observe whether the vitrification does modify their spatial distribution. To analyze this staining, we will use quantitative image analysis method.
Analysis of maternal factor stabilities. | at day 1
  Maternal factors stored in the oocyte cytoplasm during oogenesis as proteins and transcripts are essential for the early embryonic development. To know if the stock of maternal factors is diminished by the vitrification procedure, we will perform Reverse Transcription combined with Real Time PCR to quantify transcript amounts of candidates genes selected from human oocytes databases.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France